CLINICAL TRIAL: NCT03633474
Title: Lactamica 7: Defining the Immune Response to Nasopharyngeal Colonisation by the Commensal Neisseria Lactamica
Brief Title: Defining the Immune Response to Nasopharyngeal Colonisation by the Commensal Neisseria Lactamica
Acronym: Lac-7
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Lactamica-7
Record Dates: First submitted 2018-08-13; First posted 2018-08-16 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Meningitis, Bacterial
Keywords: Healthy volunteer; Human Challenge study
MeSH Terms: conditions — Meningitis, Bacterial

STUDY DESIGN:
Intervention Model Description: Volunteers will be blinded to the inoculum type received (i.e. N. lactamica or PBS control) throughout the study duration. Nasal secretion and throat swabs will be taken to enable mucosal immune profiling and microbiome analyses to be performed. Subjects will be screened for nasopharyngeal N. meningitidis carriage -28 to -7 days (visit 1) and non-Neisseria spp. carriers will be challenged with either 105 cfu N. lactamica suspended in PBS or PBS only control (day 0, visit 2). Volunteers identified as carriers of N. meningitidis at visit 1 will be excluded from the study and will not progress to experimental human challenge. Biological samples (nasal secretion, microbiome swab and blood) will be collected from volunteers who progress to the challenge (visit 2, Day 0) and on days +7 (+/-3), +14 (+/-3) and +28 (+/-5) post-challenge. Nasal wash sampling will not be taken at the challenge visit (Day 0) but will be taken on days +7(+/-3), +14 (+/-3) and +28 (+/-5) post-challenge.
Who Masked: Participant
Masking Description: Non-Neisseria spp. carriers will randomised in a ratio of 2:1 to receive either 10-5 cfu N. lactamica or PBS control using randomisation software, e.g. Sealed envelope (TM) available online.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- N. Lactamica in PBS (Experimental): Wild-type Neisseria lactamica (strain Y92-1009, sequence type 3493, clonal complex 613) will be used for this human challenge experiment. This strain is identical to that utilised in our previous challenge experiments (>350 volunteers to date).
  Interventions: Biological: N. lactamica
- PBS Control (Placebo Comparator): PBS only control. Volunteers randomized to this arm will receive a PBS only solution which contains no bacteria.
  Interventions: Other: PBS only

INTERVENTIONS:
Biological: N. lactamica — Stocks of N. lactamica (strain Y92-1009, sequence type 3493, clonal complex 613) in Frantz medium containing 30% (v/v) glycerol have been previously prepared using the Good Manufacturing Practices pharmaceutical manufacturing facilities at Public Health England (Porton Down, United Kingdom).
  Arms: N. Lactamica in PBS
Other: PBS only — Sterile PBS only containing no bacteria
  Arms: PBS Control

SUMMARY:
Neisseria meningitidis is a 'bad bacteria' which lives harmlessly in the nose and throat of many young adults (a process called colonisation). However, it can occasionally cause serious disease including meningitis. Vaccines have proven effective in preventing disease associated with a number of strains of this bacterium, however some disease-causing strains are not covered by currently available vaccines. This research is focused on exploring new approaches to preventing colonisation and disease caused by this bacterium.

Neisseria lactamica is a 'good bacteria' that colonises the nose and throat of young children. It does not cause disease in healthy people. In a previous study it has been demonstrated that the introduction of Neisseria lactamica into the noses of healthy adult volunteers resulted in a significant decrease in Neisseria meningitidis colonisation. However, it is not yet understood why this effect occurs. One theory is that the immune response the body mounts in response to colonisation with the 'good bacteria' cross-reacts with the 'bad bacteria' and in so doing eradicates the bad bacteria from the nose and throat. This study aims to outline the nature of the immune responses mounted in response to colonisation with the good bacteria, N. lactamica, after introducing it into the noses of healthy adult volunteers. In addition, the study aims to establish how the introduction of the good bacteria changes the other bacterial populations that live in the nose and throat.

DETAILED DESCRIPTION:
The clinical trial is a controlled, volunteer blinded, N. lactamica human challenge study to enable N. lactamica-specific cellular immune responses to be outlined in detail. In addition, The aim is to determine whether responses directed towards N. lactamica are cross-reactive with N. meningitidis.

Following enrolment onto the study, non-meningococcal carriers (as determined by microbiological culture of nasopharyngeal wash and retropharyngeal swab) will be challenged intra-nasally with either 10-5 cfu of N. lactamica wild-type strain Y92-1009 (30,31) suspended in sterile phosphate buffered saline (PBS), as used in previous studies, or PBS alone (control group).

Following inoculation on Day 0, biological samples (nasal wash, nasal secretion, throat swabs and blood) will be taken from all volunteers on days +7 (+/-3), +14(+/-3) and +28(+/-5) post-challenge. On the day of inoculation (Day 0) the biological samples listed will be taken except for the nasal wash.

N. lactamica-specific B-cell and CD4+ memory T-cell responses will be measured in blood using a selection of in vitro assays and the results compared longitudinally in N. lactamica challenged (colonised or non-colonised) vs. control challenged subjects. The experiments will establish the nature of T-cell and B-cell memory responses and plasma B-cell responses induced in response to N. lactamica colonisation and will determine if these responses are cross-reactive with N. meningitidis. Mucosal immune profiling and microbiome analyses will be performed on nasal secretion and nasal bacterial samples, respectively. Any remaining biological samples (following experiments performed to meet the current study objectives) will be transferred to our registered human tissue bank to enable future studies following additional ethics approval by the relevant bodies.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 18 to 45 years inclusive on the day of enrolment.
* Fully conversant in the English language.
* Able and willing (in the investigator's opinion) to comply with all study requirements.
* Written informed consent to participate in the study.
* For females only, willingness to practice continuous effective contraception (see below) during the study and negative pregnancy test at visit 1 (screening).

Exclusion Criteria:

* Active smokers.
* N. meningitidis or N. lactamica detected following culture of throat swab or nasal wash taken before the challenge.
* Individuals who have a current infection at the time of inoculation.
* Individuals who have been involved in other clinical studies/trials involving receipt of an investigational product over the last 12 weeks or if there is planned use of an investigational product during the study period.
* Individuals who have previously been involved in clinical studies/trials investigating meningococcal vaccines or experimental challenge with N. lactamica.
* Use of oral or intravenous antibiotics within the period 30 days prior to the challenge.
* Any confirmed or suspected immunosuppressive or immunocompromised state, including HIV infection, asplenia, history of recurrent severe infections or use (more than 14 days) of immunosuppressant medication within the past 6 months (topical/inhaled steroids are allowed).
* Use of immunoglobulins or blood products within 3 months prior to enrolment.
* History of blood donation within the past 12 weeks for male volunteers, or 16 weeks for female volunteers.
* Allergy to yeast extract.
* Any other significant disease, disorder, or finding which may significantly increase the risk to the volunteer because of participation in the study, affect the ability of the volunteer to participate in the study, or impair interpretation of the study data, for example recent surgery to the nasopharynx.
* Occupational, household or intimate contact with immunosuppressed persons.
* Pregnancy or lactation.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
To measure host T-cell and B-cell memory responses and plasma B-cell responses in blood to experimentally-induced nasopharyngeal colonisation with N. lactamica. | Up to Day 33
  Measurements from baseline will compare the host T and B-cell memory response (ug/mL) to samples taken post inoculation.

SECONDARY OUTCOMES:
Determine if N. lactamica-specific CD4+ T-cell memory responses detected in blood cross-react with N. meningitidis. | Up to Day 33
  From PBMC isolation of participants blood, measure if the T-cell response reacts when presented with N. meningitidis (ug/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Adam P Dale, Principal Investigator — University of Southampton
Locations (1):
- NIHR Southampton Clinical Research Facility, Southampton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dale AP, Theodosiou AA, Gbesemete DF, Guy JM, Jones EF, Hill AR, Ibrahim MM, de Graaf H, Ahmed M, Faust SN, Gorringe AR, Polak ME, Laver JR, Read RC. Effect of colonisation with Neisseria lactamica on cross-reactive anti-meningococcal B-cell responses: a randomised, controlled, human infection trial. Lancet Microbe. 2022 Dec;3(12):e931-e943. doi: 10.1016/S2666-5247(22)00283-X. PMID 36462524